CLINICAL TRIAL: NCT07077564
Title: A Single-Center, Single-Arm, Phase II Clinical Trial of TROP2-ADC in Patients With Advanced Extrapulmonary High-Grade Neuroendocrine Tumors Refractory to Standard Therapy
Brief Title: The Efficacy of TROP2-ADC in Advanced Extrapulmonary High-Grade Neuroendocrine Neoplasms Failure of Standard Therapy
Acronym: SKB264-II-NEN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0615
Record Dates: First submitted 2025-07-10; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Neuroendocrine Neoplasms (Tumours)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab govitecan 5 mg/kg every 2 weeks on Day 1 of each cycle（iv） (Experimental)
  Interventions: Drug: Sac-TMT

INTERVENTIONS:
Drug: Sac-TMT — Sacituzumab govitecan 5 mg/kg every 2 weeks on Day 1 of each cycle（IV）

SUMMARY:
The response rate to second-line or later therapies for extrapulmonary high-grade neuroendocrine neoplasms (NENs) remains low, with no established standard treatment regimen. Patients exhibit short survival periods, with median overall survival ranging from 5.1 to 18 months, representing a significant unmet clinical need. Sacituzumab govitecan has been evaluated in multiple clinical trials including OptiTROP-Breast01, KL264-01, OptiTROP-Lung01, OptiTROP-Lung03, and SKB264-Ⅱ-06. Current results consistently indicate promising efficacy of Sacituzumab govitecan in lung cancer, breast cancer, and cervical cancer. Notably, data presented at the 2025 American Society of Clinical Oncology (ASCO) Annual Meeting revealed that TROP2 is highly expressed in neuroendocrine tumors, and its expression is significantly associated with poor prognosis. This suggests TROP2-directed antibody-drug conjugates (ADCs) may demonstrate promising therapeutic potential in NENs.

Research Objective:To evaluate the efficacy of Sacituzumab govitecan in patients with advanced extrapulmonary neuroendocrine neoplasms who have progressed on standard therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and voluntarily participate in the study.
2. Aged 18-75 years, male or female.
3. Histologically or cytologically confirmed diagnosis of one of the following:

   Metastatic neuroendocrine carcinoma (NEC) Neuroendocrine tumor (NET) Grade 3 (G3) Mixed neuroendocrine-non-neuroendocrine neoplasm (MiNEN) with >30% neuroendocrine component.
4. Progression after at least one prior line of systemic therapy.
5. ECOG Performance Status of 0 or 1.
6. Life expectancy ≥3 months.
7. At least one measurable lesion per RECIST 1.1 at baseline:
8. Lesions must not have received prior local therapy (e.g., radiotherapy). Lesions within prior radiotherapy fields are acceptable if progression is documented.
9. Adequate organ function (no blood products/growth factors within 14 days prior):

   * Absolute neutrophil count (ANC) ≥1.5×10⁹/L

     * Platelets ≥100×10⁹/L ③Hemoglobin ≥8 g/dL ④Total bilirubin ≤1.5 × ULN ⑤ALT/AST ≤2.5 × ULN (≤5 × ULN if liver metastases present) ⑥Serum creatinine ≤1.5 × ULN or creatinine clearance >60 mL/min (Cockcroft-Gault formula).

9. Contraception requirements:

Females of childbearing potential:

Negative serum pregnancy test within 72 hours prior to dosing. Use highly effective contraception (e.g., IUD, oral contraceptives, condoms) during and for ≥3 months after last dose.

Males with fertile partners:

Use effective contraception during and for ≥3 months after last dose.

Exclusion Criteria:

* (1) Active CNS metastases and/or carcinomatous meningitis.

  * Exception: Subjects with treated brain metastases may enroll if: Stable for ≥28 days prior to study initiation, Off steroids for brain metastases ≥28 days. Note: Carcinomatous meningitis excluded regardless of stability.

    (2) Major surgery, open biopsy, or significant trauma within 28 days prior to first dose.

    (3) History of severe interstitial lung disease (ILD) with inadequate control. (4) Uncontrolled hypertension (SBP ≥140 mmHg or DBP ≥90 mmHg despite antihypertensive therapy).

    (5) Poorly controlled cardiovascular disease, including:
    1. NYHA Class II+ heart failure
    2. Unstable angina
    3. Myocardial infarction within 1 year
    4. Clinically significant supraventricular/ventricular arrhythmias refractory to intervention (6) Clinically significant bleeding within 3 months prior to first dose (e.g., GI bleeding, hemorrhagic gastric ulcer, vasculitis). (7) Arterial/venous thromboembolic events within 6 months prior to first dose (e.g., CVA, TIA, cerebral hemorrhage, DVT, PE).Exception: Superficial thrombosis per investigator assessment.

       (8) Active other malignancy requiring therapy. Exceptions: Non-melanoma skin cancer in situ with curative treatment.

       (9)Pregnancy or lactation. (10)Other factors potentially leading to premature discontinuation per investigator judgment: Severe comorbidities (including psychiatric), Critical lab abnormalities, Social/familial factors compromising safety/data integrity (11)TROP2-targeted agents, ADC drugs (e.g., 8201)Topoisomerase I inhibitor-containing ADCs (12)Live vaccination within 30 days prior to first dose or planned during study.

       (13)Requirement for strong CYP3A4 inhibitors/inducers within 2 weeks prior to first dose or during study.

       (14) Palliative radiotherapy to known metastatic sites within 2 weeks prior to first dose.

       (15)Systemic anti-infective therapy within 1 week prior to first dose. Severe ocular conditions including: (16)Dry eye syndrome, Meibomian gland dysfunction, Blepharitis, Corneal disease delaying healing (17)Other exclusionary conditions per investigator assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2028-07-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | 2 months
  The proportion of patients whose tumor volume has decreased to a pre-specified value (CR/PR) according to RECIST version 1.1 for solid tumors and can maintain the minimum required duration.

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | 2 years
  Refers to the time from the start of randomization (or the start of treatment in a single-arm trial) until tumor progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | 2 years
  The proportion of patients with solid tumors (according to RECIST version 1.1) who achieve remission (PR+CR) and stable disease (SD) after treatment and can maintain the minimum required duration.
Overall Survival(OS) | 2 years
  Refers to the time from the start of randomization (or the start of treatment in a single-arm trial) until death due to any cause.

OTHER OUTCOMES:
Adverse Event (AE) | 2 years
  In a drug clinical trial, it refers to all adverse medical events that occur in subjects after receiving the investigational medicinal product, which can manifest as symptoms, signs, diseases, or laboratory abnormalities, but are not necessarily causally related to the investigational medicinal product.